CLINICAL TRIAL: NCT05158842
Title: Optimising the Treatment of COVID-19 Positive/Negative Adults With Severe Pneumonia and/or ARDS in Bangladesh Using an Adaptive Version of Locally Made Bubble CPAP: Feasibility Study
Brief Title: Treatment of COVID-19 Positive/Negative Bangladeshi Adults With Severe Respiratory Complaints by a Locally Made bCPAP: Feasibility Study
Acronym: Adult-bCPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Dhaka Medical College (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PR-20065
Record Dates: First submitted 2021-03-29; First posted 2021-12-15 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-02

CONDITIONS: Severe Pneumonia; Acute Respiratory Distress Syndrome; Covid19
Keywords: Feasibility; COVID-19; Bubble CPAP; Acute Respiratory Distress Syndrome; Severe Pneumonia
MeSH Terms: conditions — Pneumonia; Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bubble CPAP Oxygen Therapy (Other): Feasibility of Device
  Interventions: Device: Adult bubble CPAP oxygen therapy device

INTERVENTIONS:
Device: Adult bubble CPAP oxygen therapy device — In Bubble CPAP, pressurized oxygen from an oxygen cylinder is delivered to the patient. Adjusting the height of the water column above the exit of the tube can regulate the pressure in the system and the amount of CPAP delivered to the patient. Oxygen is delivered by a successfully tested, silicon-based, ergonomically designed adaptive version of nasal canula (nasal seal) inserted into the nostril of a patient.
  The components are:
  1. Adaptive version of nasal canula (nasal seal)
  2. A nasal canula with connecting circuit system
  3. Water-filled bottle with marking water pressure from10 to15 L/min.
  Oxygen cylinder, central distribution through pipelines or by oxygen concentrator will be used as an oxygen source.

SUMMARY:
Low and middle-income countries (LMICs) urgently need cost-effective adaptive technologies to provide CPAP. The lead investigator has designed a device that has already been approved by the Directorate General of Drug Administration (DGDA), Government of the People's Republic of Bangladesh.

The design of the nasal seal was comfortable and well tolerated by all the participants. Patients were told about some mild discomfort at higher delivered pressures (14 or 15 cm PEEP), consistent with pressurised nasal delivery by similar devices.

The safety phase has been initiated since 1st November 2020 and ended in April 2021. One patient withdrew from the study but none of them developed any adverse events.

The feasibility phase started at the end of September 2021.

Objectives:

1. To evaluate the barriers and operational challenges related to the introduction of adult bubble CPAP oxygen therapy
2. To evaluate the acceptability of introducing adult bubble CPAP in tertiary level hospitals of Bangladesh

DETAILED DESCRIPTION:
Low and middle-income countries (LMICs) urgently need cost-effective adaptive technologies to provide CPAP. The lead investigator has proved that a low cost, locally made bCPAP device is capable of reducing mortality in children, Its components are (a) an interface; nasal seal, (b) oxygen delivery piping, connectors and nasal cannula, (c) appropriately sized transparent plastic bottles (containing sterilized water). The device and its components are already being approved by the Directorate General of Drug Administration (DGDA), Government of the People's Republic of Bangladesh. Adapting this technology, if safe and scaled up, could possibly decrease the need for mechanical ventilation and subsequently averting deaths among adult COVID-19 patients.

The design of the nasal seal was comfortable and well tolerated by all the participants. Patients were told about some mild discomfort at higher delivered pressures (14 or 15 cm PEEP), consistent with pressurised nasal delivery by similar devices. No additional adverse events such as trauma/injury, erosion, bruise, bleeding, obstruction, breathlessness, pneumothorax, pneumomediastinum, abdominal distension during and after the trial were reported.

The safety phase has been initiated since 1st November 2020 and ended in April 2021. One patient withdrew from the study but none of them developed any adverse events.

The feasibility phase started at the end of September 2021.

Objectives:

1. To evaluate the barriers and operational challenges related to the introduction of adult bubble CPAP oxygen therapy
2. To evaluate the acceptability of introducing adult bubble CPAP in tertiary level hospitals of Bangladesh

ELIGIBILITY:
INCLUSION CRITERIA

Adults for assessment:

* Male or female
* RT-PCR positive or negative for COVID-19
* Aged 18-64 years, with severe pneumonia and hypoxemia (SpO2 < 90%).
* Willing and able to provide written informed consent.

Staff:

* Staff (physicians and nurses) who are engaged in the medicine ward, HDU and COVID ward of Dhaka Hospital of icddr,b and Dhaka Medical College Hospital.
* Staff who agree to participate and give written informed consent.

EXCLUSION CRITERIA

Adults for assessment:

* Patients will not be included in the study if they will not have adequate respiratory drive such as gasping respiration or requiring cardiopulmonary resuscitation or
* Known to have life threatening heart disease,
* Status asthmaticus
* Upper-airway obstruction
* Patients with pneumonia/respiratory tract illness but without hypoxaemia or SpO2< 80% in room air even on prone position and chest physiotherapy
* Pregnancy, nasal polyp and
* Patients who are not willing or able to provide written informed consent.
* Arterial blood gas analysis will be performed to check the exclusion criteria.

Staff:

• For Focus Group Discussions, physicians and nurses who do not provide written informed consent will be excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Optimising the treatment of COVID-19 positive/negative adults with severe pneumonia and/or ARDS in Bangladesh using an adaptive version of locally made Bubble CPAP: Feasibility study | 17 weeks
  Barriers and operational challenges related to the introduction of adult bubble CPAP oxygen therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammod J Chisti, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (2):
- Bangladesh (2):
  - Dhaka Hospital, ICDDR,B, Dhaka
  - Dhaka Medical College Hospital, Dhaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO. Clinical management of severe acute respiratory infection (SARI) when COVID-19 disease is suspected. Interim guidance, 13 March 2020. 2020 [1-21]
- [Result] Chisti MJ, Salam MA, Smith JH, Ahmed T, Pietroni MA, Shahunja KM, Shahid AS, Faruque AS, Ashraf H, Bardhan PK, Sharifuzzaman, Graham SM, Duke T. Bubble continuous positive airway pressure for children with severe pneumonia and hypoxaemia in Bangladesh: an open, randomised controlled trial. Lancet. 2015 Sep 12;386(9998):1057-65. doi: 10.1016/S0140-6736(15)60249-5. Epub 2015 Aug 19. PMID 26296950